CLINICAL TRIAL: NCT01870024
Title: Comparison Between Lorazepam, Clonazepam and Clonazepam + Fosphenytoin for the Treatment of Out-of-hospital Generalized Status Epilepticus in Adults Patients
Brief Title: Comparison Between Lorazepam, Clonazepam and Clonazepam + Fosphenytoin for the Treatment of Out-of-hospital Generalized Status Epilepticus
Acronym: LORACLOFT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P110123; 2012-003795-39 (EudraCT Number)
Record Dates: First submitted 2013-06-03; First posted 2013-06-05 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Status Epilepticus; Epilepsy
Keywords: status epilepticus; epilepsy; seizures; convulsive seizures; convulsions; benzodiazepines; anticonvulsants
MeSH Terms: conditions — Status Epilepticus; Epilepsy; Seizures | interventions — Clonazepam; fosphenytoin; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1: Lorazepam + Placebo (Active Comparator): [ L + P ] = lorazepam 0,1mg/kg by intravenous injection over a period of 2 to 3 minutes) + placebo 20 mg/kg by intravenous infusion over a period of 15 minutes
  Interventions: Drug: Placebo; Drug: Lorazepam
- 2: Clonazepam + Placebo (Active Comparator): [ C + P ] = clonazepam 0,015 mg/kg by intravenous injection over a period of 2 to 3 minutes + placebo 20 mg/kg by intravenous infusion over a period of 2 15 minutes
  Interventions: Drug: Clonazepam; Drug: Placebo
- 3: Clonazepam + Fosphenytoin (Active Comparator): [ C + F ] = clonazepam 0,015 mg/kg by intravenous injection over a period of 2 to 3 minutes + fosphenytoin 20 mg/kg Equivalent Phenytoin (EP) by intravenous infusion over a period of 15 minutes
  Interventions: Drug: Clonazepam; Drug: Fosphenytoin

INTERVENTIONS:
Drug: Clonazepam — clonazepam 0,015 mg/kg
  Arms: 2: Clonazepam + Placebo; 3: Clonazepam + Fosphenytoin
Drug: Fosphenytoin — fosphenytoin 20 mg/kg Equivalent Phenytoin (EP) by intravenous infusion over a period of 15 minutes
  Arms: 3: Clonazepam + Fosphenytoin
Drug: Placebo — placebo 20 mg/kg by intravenous infusion over a period of 15 minutes
  Arms: 1: Lorazepam + Placebo; 2: Clonazepam + Placebo
Drug: Lorazepam — lorazepam 0,1mg/kg by intravenous injection over a period of 2 to 3 minutes)
  Arms: 1: Lorazepam + Placebo

SUMMARY:
The main purpose of this study is to know on one hand if lorazepam is more (effective) than clonazepam and on the other hand if lorazepam is also effective as the association clonazepam + fosphenytoin in out-of-hospital treatment of the generalized convulsive status epilepticus in adult patients.

DETAILED DESCRIPTION:
Background: Early and rapid termination of status epilepticus with intravenous administration of benzodiazepines only or its association with other antiepileptic drug improves outcomes. Our out-of-hospital study aims to demonstrate on one hand the superiority of lorazepam compared with clonazepam and on the other hand the efficacy at least equivalent of lorazepam in comparison with the association clonazepam + fosphenytoin. If these hypotheses are demonstrated, the out-of-hospital treatment of the status epilepticus by lorazepam in monotherapy would then be strongly recommended, considering its efficacy and the simplicity of administration in the context of the pre-hospital emergency.Objective: To compare the efficacy of Lorazepam with that of Clonazepam and its association with Fosphenytoin for the treatment of out-of-hospital status epilepticus.

Participating centers: 41 prehospital emergency services employing mobile intensive care units and located in urban areas in France participated in this study. In France, the management of out-of-hospital medical emergencies is under the responsibility of the Service d'Aide Medicale Urgente (SAMU). Mobile intensive care units are staffed by an attending emergency physician or anesthesiologist, a nurse, and an ambulance driver. The study is coordinated by the prehospital emergency service of Lariboisiere Hospital, University Paris 7 (Paris, France)

Number of patients: 522 patients; 174 patients by group.

Duration of the study: The total duration planned is of 48 months Intermediate analysis: An intermediate analysis is planned while 261 patients will be included (50 % of the inclusions).Duration of participation of every patient: 24 hours Data collection: prehospital data recording during the 60 min period of the study, and intrahospital data recording by the medical report of hospitalization.

Methodology: Multicenter, randomized, double-blind trial with 3 arms.

Main criteria of evaluation: the cessation of the status epilepticus and the absence of recurrence from T20 minutes until T60 minutes after the beginning of the treatment.

The cessation of the status epilepticus is defined by the stop of any motor activity and any seizures or convulsive movements. The absence of recurrence is defined by the not occurrence of a new seizures after a period of cessation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Out-of-hospital management
* presenting one of the criteria below noticed by the physician of the mobile intensive care unit:

  1. convulsive seizures at the time of treatment and were reported by reliable witnesses to have been continuously convulsing for longer than 5 minutes, without regaining consciousness, or
  2. if they were having more than 2 repeated convulsive seizures at the time of treatment without regaining consciousness

Exclusion Criteria:

* Patient having been already included in the study during a previous episode of status epilepticus
* Patient having already received before the arrival of the mobile intensive care unit one of theses studied drugs (lorazepam, clonazepam or fosphenytoin or phenytoin)
* Latent status epilepticus in deep coma
* Cerebral anoxia (post cardio respiratory arrest)
* Severe head trauma
* Patient presenting convulsive seizures of psychogenic origin
* Lennox Gastaut's syndrome
* Decision of urgent intubation
* Patients of more than 110 kg ( estimated weight
* Heart rate < 60 bpm or > 150 bpm
* Systolic Blood Pressure < 90 mmHg
* Atrioventricular block of 2nd or 3rd degree
* Ventricular tachycardia or ventricular fibrillation
* Sensibility known about benzodiazepines, fosphenytoin, phenytoin, other hydantoins, or barbiturate
* Contraindication known about benzodiazepines (severe respiratory failure, severe acute hepatic failure, myasthenia, syndrome of sleep apnea, glaucoma with closed angle
* Contraindication known about fosphenytoin (intermittent acute porphyry)
* Contraindication known about barbiturate (porphyry, severe respiratory failure, current treatment by saquinavir, ifosfamide and voriconazole, in association with millepertuis)
* Person unaffiliated in a National Social Security Insurance
* Pregnant or breast-feeding Woman
* Impossibility to put an intravenous or intra-osseous catheter for the treatment injection
* Absence of nurse in the mobile intensive care unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 434 (Actual)
Dates: Start 2013-06-26 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Percentage of patient with a cessation of seizures and absence of recurrence | between 20 and 60 minutes after the beginning of the treatment
  Percentage of patient with a cessation of seizures and absence of recurrence from 20 minutes until 60 minutes after the beginning of the treatment

SECONDARY OUTCOMES:
Duration between the first cessation and the recurrence of seizures | up to 60 minutes
  Duration between the first cessation and the recurrence of seizures
Percentage of patients having had a second injection of benzodiazepine | up to 60 minutes
  Percentage of patients having had a second injection of benzodiazepine
Percentage of patients having had an injection of the second line treatment | up to 60 minutes
  Percentage of patients having had an injection of the second line treatment (i.e. Fosphenytoin or barbiturate)
Percentage of patients having a general anesthesia for refractory status epilepticus | up to 60 minutes
  Percentage of patients having a general anesthesia for refractory status epilepticus
Percentage of patients having had a side effect | up to 60 minutes
  Percentage of patients having had a side effect (low blood pressure, arrhythmias)
Percentage of patients having been mechanically ventilated | up to 60 minutes
  Percentage of patients having been mechanically ventilated in pre-hospital setting
Glasgow Coma Scale | 60 minutes
  Glasgow Coma Scale on arrival at the hospital
Mortality | up to 60 minutes
  Mortality in pre-hospital setting
Mortality | up to Day 30
  Mortality in hospital until J30 (if the patient still hospitalized)
Length of stay in Intensive Care Unit | up to Day 30
  Length of stay in Intensive Care Unit
Length of stay in hospital | up to Day 30
  Length of stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Papa GUEYE, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris; François CONCINA, MD, Principal Investigator — CHU Toulouse - Hôpital Purpan
Locations (1):
- Département d'Anesthésie - Réanimation - SMUR - Hôpital Lariboisière, Paris, France